CLINICAL TRIAL: NCT06721130
Title: Role of 18F-FDG PET/CT in the Evaluation of Cavernous Sinus Syndrome: a Pilot Study
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Rajender Kumar, Additional Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Other Study IDs: 1134
Record Dates: First submitted 2024-11-27; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2022-07

CONDITIONS: Cavernous Sinus Syndrome; Cavernous Sinus Meningioma; Cavernous Sinus Lesions
Keywords: Cavernous Sinus Syndromes; Ophthalmoplegia; Positron Emission Tomography Computed Tomography; Fluorodeoxyglucose F18; Cavernous Sinus
MeSH Terms: conditions — Cavernous Sinus Syndromes; Ophthalmoplegia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Treatment naive patients presenting with Cavernous Sinus Syndrome with cavernous sinus lesion on MRI
  Interventions: Diagnostic Test: FDG radiotracer

INTERVENTIONS:
Diagnostic Test: FDG radiotracer — Pilot study evaluating the role of FDG PET/CT in Cavernous sinus syndrome
  Other Names: FDG PET/CT

SUMMARY:
Cavernous sinus syndrome (CSS) can be caused by a wide range of inflammatory, malignant, benign, vascular and miscellaneous disorders. Even after modern advances, reaching the final etiological diagnosis remains a challenge in CSS. This study is planned to determine the role and incremental value of 18F-FDG PET/CT in characterising different cavernous sinus pathologies based on their metabolic activity and detecting extracranial involvement.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age greater than or equal to 18 years,
2. with newly diagnosed CSS,
3. lesion seen on MRI in the CS, and
4. willing to give written informed consent.

Exclusion Criteria:

1. Pregnant and lactating patients
2. Patients already being treated (including steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive treatment naive patients of either sex with signs and symptoms of cavernous sinus syndrome attending the outpatient clinic in the Department of Neurology, Postgraduate Institute of medical Education & Research, Chandigarh.
  Case definition for CSS- involvement of two or more cranial nerves (which pass through CS) or oculosympathetic fibers on the same side, or involvement of only cranial nerve in combination with a radiologically confirmed cavernous sinus lesion.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
SUVmax of the cavernous sinus lesions on FDG PET/CT | From enrollment to the establishment of final diagnosis upto a period of three months
  Standardized uptake value (SUV) will be calculated by drawing region of interest (ROI) in the cavernous sinus region both on the whole body and the dedicated brain image, while carefully excluding normal brain activity. If lesions in the bilateral cavernous sinuses will be present, SUVmax of both the lesions will be noted.
Number of patients with extracranial sites of involvement on FDG PET/CT | From enrollment to the establishment of final diagnosis upto 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India